CLINICAL TRIAL: NCT07085663
Title: Exergame-assisted Simultaneous Motor-cognitive Training for Middle-aged Old Adults in China: a Feasibility and Pilot Randomized Controlled Trail Study
Brief Title: Exergame-assisted Simultaneous Motor-cognitive Training for Middle-aged Old Adults in China
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Principal Investigator, LI Yaqin, Principal Investigator, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HSEARS20240516005
Record Dates: First submitted 2025-05-08; First posted 2025-07-25 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Subjective Cognitive Decline
Keywords: exergame; subjective cognitive decline; middle-aged; physical performance; cognitive performance; dual-task performance

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exergame-assisted motor-cognitive training group (Experimental): Exergame-assisted motor-cognitive training group
  Interventions: Other: Exergame-assisted simultaneous motor-cognitive training
- Blank control (No Intervention): Blank control

INTERVENTIONS:
Other: Exergame-assisted simultaneous motor-cognitive training — Exergame-assisted simultaneous motor-cognitive training
  Arms: Exergame-assisted motor-cognitive training group

SUMMARY:
To develop and conduct a pilot trial on the effectiveness of a technology-based (exergame) intervention approach for the middle-aged old adults' population in China. The study will examine the feasibility of the intervention and estimate its preliminary effects in improving their physical, cognitive, and dual-task performance.

ELIGIBILITY:
Inclusion Criteria:

* people between 50 and 60 years of age
* living in mainland China
* confirmed subjective cognitive decline with the following diagnostic criteria; a confirmed case of subjective cognitive decline that meets the subjective cognitive decline-9 scale and an exclusion of mild cognitive impairment cases using the Montreal Cognitive Assessment scale to rule out mild cognitive impairment; subjective decline in memory rather than other cognitive domains; episodes of subjective cognitive decline within the past 5 years; participants perceived to experience a sustained decline in cognitive performance compared to previous normality, independent of an acute event.
* the absence of a medical condition that renders exercise inappropriate. This includes, but is not limited to, heart disease, hypertension, diabetes, respiratory disease (e.g., chronic obstructive pulmonary disease), joint and bone disease, and neurological disease (e.g., parkinson's disease)
* have the ability to perform independent activities of daily living (as measured by the independent activities of daily living scale)
* have no history of falls
* have no language barriers and have adequate communication skills

Exclusion Criteria:

* active mental disorder, serious mental illness, neurological disorder, or cognitive impairment (standard mild cognitive impairment, prodromal Alzheimer's disease or dementia, or other significant cognitive deficits)
* substance use for a long-term mental or neurological illness
* severe mobility or sensory impairments that may prevent participation in research activities
* unstable or acute medical conditions
* individuals who have recently undergone major surgery or have acute orthopedic conditions
* individuals who refuse to participate

Ages: 50 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-05-20 (Actual); Primary Completion 2025-08-30 (Estimated); Study Completion 2025-08-30 (Estimated)

PRIMARY OUTCOMES:
Recruitment rate of the exergame-assisted simultaneous motor-cognitive training (percentage) | From "recruiment" and "immediately after the completion" (no follow-up, intervention duration-4 weeks)
  Recruitment rate = (number of successful applicants ÷ total number of potential applicants) × 100%. The higher the percentage, the better the recruitment efficiency.The recruitment rate is calculated after the experiment ends, with all potential participants and successful participants recorded throughout the process.
Retention rate of the exergame-assisted simultaneous motor-cognitive training (percentage) | From "recruiment" and "immediately after the completion" (no follow-up, intervention duration-4 weeks)
  Retention rate = (number of participants still employed at the end of the experiment ÷ number of participants employed at the beginning of the experiment) × 100%. The higher the ratio, the better feasibility.The retention rate is calculated after the experiment ends, with recording of all participants still employed and participants employed at the beginning of the experiment throughout the whole process.
Adherence of the exergame-assisted simultaneous motor-cognitive training (percentage) | From "recruiment" and "immediately after the completion" (no follow-up, intervention duration-4 weeks)
  Adherence = (actual number of interventions completed ÷ total number of planned interventions) × 100%. Adherence ≥80% indicates good intervention feasibility (supporting formal RCT implementation), <70% suggests that the programme needs to be optimised (e.g. adjusting intensity, frequency or support measures), and if the adherence rate for key steps (e.g. medication) is <50%, this may affect the validity assessment.
Acceptability of the exergame-assisted simultaneous motor-cognitive training (narrative description) | From "recruiment" and "immediately after the completion" (no follow-up, intervention duration-4 weeks)
  The acceptability of this study will be evaluated by recording participants' evaluations of the experiment and positive/neutral/negative descriptions using a dedicated form. The more positive descriptions there will be, the better the acceptability.
Adverse events of the exergame-assisted simultaneous motor-cognitive training (narrative description) | From "recruiment" and "immediately after the completion" (no follow-up, intervention duration-4 weeks)
  The adverse events of this study will be recorded using a dedicated form (time, location, first aid treatment, causal analysis, follow-up). Adverse events are recorded throughout the entire experimental process. The less adverse events descriptions there will be, the better the feasibility

SECONDARY OUTCOMES:
Change from baseline in "grip strength" at four weeks through grip dynamometer assessment（kilograms) | From "baseline" to "immediately after the completion" (no follow-up, intervention duration-4 weeks)
  When measuring with an electronic dynamometer, the value may range from 0 (worst result) to any possible positive value (best result). Two assessment points, from "baseline" to "immediately after the completion" (no follow-up, intervention duration-4 weeks)
Change from baseline in "lower limb muscle strength and functional muscle endurance" at four weeks through "30-second chair stand"(frequency) | From "baseline" to "immediately after the completion" (no follow-up, intervention duration-4 weeks)
  Participants crossed their arms across their chest and performed the complete movement of 'fully lifting their back off the chair back → standing straight → sitting back down' as many times as possible within 30 seconds. The counting standard was that the next standing movement could only begin after the buttocks made contact with the chair seat. The assessment criteria are as follows for the 50-59 age group: males (poor: <15 times, moderate: 15-20 times, good: >20 times); for females (poor: <13 times, moderate: 13-18 times, good: >18 times). Two assessment points, from "baseline" to "immediately after the completion" (no follow-up, intervention duration-4 weeks)
Change from baseline in "lower limb muscle strength and functional muscle endurance" at four weeks through "30- second deep squat elastic band"(frequency) | From "baseline" to "immediately after the completion" (no follow-up, intervention duration-4 weeks)
  Participants stand with both feet on the middle section of the resistance band (the stength of resistance band is 20 pounds in this study), holding the band with both hands and securing it at shoulder level. Within 30 seconds, they perform as many full-range squats as possible (with thighs below the horizontal line), maintaining a straight back and knees aligned with the toes throughout the movement. The number of repetitions directly reflects lower limb muscle strength and dynamic stability, with a higher number indicating stronger functional strength. For individuals aged 50 to 60, males with fewer than 10 repetitions are considered weak, 10-14 repetitions are moderate, and 15 or more are strong; females with fewer than 8 repetitions are considered weak, 8-12 repetitions are moderate, and 13 or more are strong.Two assessment points, from "baseline" to "immediately after the completion" (no follow-up, intervention duration-4 weeks)
Change from baseline in "the ability to extend the trunk, hip joints, and posterior muscle groups of the lower limbs and the range of motion of the joints" at four weeks through "seated forward bending"(centimeters) | From "baseline" to "immediately after the completion" (no follow-up, intervention duration-4 weeks)
  Participants sit on the ground with legs straightened and heels together against the test box. Arms are extended forward, and the slider is slowly pushed to the farthest distance and held for 1 second. The position reached by the fingertips is measured (the sole of the foot is 0 points; values exceeding this are positive, and values not exceeding it are negative). The measurement value (in centimetres) reflects the flexibility of the lower back and hamstrings. A higher positive value indicates better flexibility (e.g., >+15 cm is excellent), while a negative value suggests stiffness and the need for stretching (e.g., <-5 cm indicates a risk of strain).Two assessment points, from "baseline" to "immediately after the completion" (no follow-up, intervention duration-4 weeks)
Change from baseline in "dynamic balance ability and postural control stability" at four weeks through "functional reach test, FRT"(centimeters) | From "baseline" to "immediately after the completion" (no follow-up, intervention duration-4 weeks)
  Participant stands upright with one arm extended forward. Without moving the feet, the maximum horizontal distance that the fingertips can be extended forward is measured (unit: centimetres). The distance value reflects dynamic balance ability. A forward extension distance of <15.2 cm indicates a significantly increased risk of falling (sensitivity 89%, specificity 79%), while healthy elderly people typically have a distance of ≥25 cm.Two assessment points, from "baseline" to "immediately after the completion" (no follow-up, intervention duration-4 weeks)
Change from baseline in "exercise endurance test" at four weeks through "6-minute walk test, 6MWT" (meters) | From "baseline" to "immediately after the completion" (no follow-up, intervention duration-4 weeks)
  Participants walked back and forth at their fastest pace on a 30-metre flat corridor for 6 minutes. The operator reported the time every minute and provided standardised encouragement (e.g., 'Keep going, only X minutes left'). Total walking distance (metres) directly reflects cardiopulmonary function and overall endurance. Healthy adults typically achieve 400-700 metres; a distance of <300 metres suggests severe heart failure or significantly increased risk of falls, while an increase of ≥70 metres indicates effective rehabilitation therapy.Two assessment points, from "baseline" to "immediately after the completion" (no follow-up, intervention duration-4 weeks)
Change from baseline in "functional mobility" at four weeks through "timed up and go,TUG" (seconds) | From "baseline" to "immediately after the completion" (no follow-up, intervention duration-4 weeks)
  Participants stand up from a chair with armrests, walk 3 metres at their usual pace, turn around, and return to sit down again. The entire process is timed (in seconds), and the use of conventional walking aids is permitted. The completion time directly reflects dynamic balance and fall risk. A time of ≥12 seconds indicates a significantly increased risk of falling (community elderly threshold value). Specific thresholds should be adjusted based on the population (e.g., ≥11.5 seconds for Parkinson's disease patients, ≥10 seconds for hip arthritis patients).Two assessment points, from "baseline" to "immediately after the completion" (no follow-up, intervention duration-4 weeks)
Change from baseline in "static balance ability" at four weeks through "one-legged standing, OLS" (seconds) | From "baseline" to "immediately after the completion" (no follow-up, intervention duration-4 weeks)
  Participants stand on one leg with their eyes open (they may choose to place their hands on their hips or let them hang naturally), with the other leg bent and lifted off the ground. The maximum time spent maintaining balance is recorded (in seconds). The testing process must be conducted with full fall prevention measures in place. Standing time reflects static balance ability. Healthy adults typically achieve ≥30 seconds (for the 30-year-old population), while <10 seconds indicates a significantly increased risk of falls (a sensitive indicator for the elderly). Specific results should be interpreted in conjunction with age-specific standards (e.g., ≥15 seconds is considered normal for those aged 60 years). Two assessment points, from "baseline" to "immediately after the completion" (no follow-up, intervention duration-4 weeks)
Change from baseline in "cognitive function" at four weeks through scale(total score) by "the Montreal Cognitive Assessment" | From "baseline" to "immediately after the completion" (no follow-up, intervention duration-4 weeks)
  Participants completed multiple cognitive domain tests included in this scale (including memory, visuospatial, executive function, attention, language, etc.), covering tasks such as alternating line drawing, cube copying, clock drawing, word recall, calculation, and orientation. The total score of the scale is 30 points. A score of ≥26 points (or ≥25 points after adjustment) indicates normal cognitive function, while a score of ≤22 points suggests mild cognitive impairment (MCI). Two assessment points, from "baseline" to "immediately after the completion" (no follow-up, intervention duration-4 weeks)
Change from baseline in "cognitive function" at four weeks through scale(total score) by "the Subjective Cognitive Decline-9" | From "baseline" to "immediately after the completion" (no follow-up, intervention duration-4 weeks)
  Participants answered nine questions about the frequency of recent declines in memory using a self-report questionnaire. Each question was scored using a two-category option (yes = 1 point, no = 0 points) or a three-category option (often = 1 point, occasionally = 0.5 points, never = 0 points). A higher total score indicates more significant subjective cognitive decline, and participants with a total score of ≥5 were identified as having subjective cognitive decline.Two assessment points, from "baseline" to "immediately after the completion" (no follow-up, intervention duration-4 weeks)
Change from baseline in "cognitive function and dual-task performance" at four weeks through scales(total score and seconds taken to answer per question) by "the COGNITIVE EXPERIMENTS STANDARD TOOLBOX" | From "baseline" to "immediately after the completion" (no follow-up, intervention duration-4 weeks)
  "The COGNITIVE EXPERIMENTS STANDARD TOOLBOX" is an online cognitive testing platform. Users load standardised cognitive testing tasks (such as executive function, working memory, etc.) via the online platform or local programme and complete an adaptive experimental process (including practice and formal testing) according to the on-screen prompts. The system automatically generates cognitive ability scores based on comprehensive indicators such as accuracy and reaction time. Two assessment points, from "baseline" to "immediately after the completion" (no follow-up, intervention duration-4 weeks)
Change from baseline in "cognitive function and dual-task performance" at four weeks through scales(total score and seconds taken to answer per question) by "the automatic scoring and timing in the exergame" | From "baseline" to "immediately after the completion" (no follow-up, intervention duration-4 weeks)
  The exergame developed for this study (a total of eight sections, each divided into beginner and advanced games) are designed to train participants' various cognitive functions (including memory, attention, and executive function). The games automatically record participants' response times and scores for each section. The total score for each section (beginner or advanced) ranges from 0 to 50 points, with higher scores being better.Two assessment points, from "baseline" to "immediately after the completion" (no follow-up, intervention duration-4 weeks)

CONTACTS AND LOCATIONS:
Locations (1):
- Sichuan Tianfu New District Huayang Street Helin Community Cognitive Care Center, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Li Y, Liu Y, Leung AY, Montayre J. Technology-Assisted Motor-Cognitive Training Among Older Adults: Rapid Systematic Review of Randomized Controlled Trials. JMIR Serious Games. 2025 Jun 3;13:e67250. doi: 10.2196/67250. PMID 40460432